CLINICAL TRIAL: NCT06589687
Title: The Patient AS EDUcator in Anesthesia: Exploring the Patients' Experience During and After Unexpected Cesarean Delivery Under Neuraxial Anesthesia to Inform Anesthetic Practice. A Prospective Patient-centred Multidisciplinary Mixed-method. (PAS-EDU-uCD-NA)
Brief Title: The Patient AS EDUcator in Anesthesia: Exploring the Patients' Experience During and After Unexpected Cesarean Delivery Under Neuraxial Anesthesia to Inform Anesthetic Practice
Acronym: PAS-EDU-uCD-NA
Status: Recruiting | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 24-08
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Psychological Well Being
Keywords: cesarean delivery; patient experience; epidural
MeSH Terms: conditions — Psychological Well-Being | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unexpected cesarean delivery under neuraxial anesthesia: Patients who have an unexpected cesarean delivery under neuraxial anesthesia.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Patients will be interviewed by the research team to learn about their experience of Cesarean delivery under neuraxial anesthetic.

SUMMARY:
This study aims to explore the patients' and providers' perspectives and inform future anesthetic practice for patients undergoing unexpected cesarean delivery (CD) under neuraxial anesthesia (NA). The consideration of patients' concerns, preferences, expectations, and suggestions may lead to enhanced patient satisfaction, compliance, and quality of care that future patients receive during unexpected CD under NA. The investigators will possibly be able to identify gaps in procedural performance that warrant further investigation during the second phase of this study which will contribute to improvement of overall patient care. During the third phase, educational material will be generated from patient insights and will be distributed to the Department of Anesthesia, Department of Obstetrics and Gynaecology, Labour and Delivery Nurses and team of Anesthesia Assistants and Respiratory Therapists.

DETAILED DESCRIPTION:
Cesarean delivery (CD) is a surgical procedure that allows for birth of a neonate through a laparotomy and hysterotomy and is the most common surgical procedure performed worldwide with 21% of all childbirths occurring via CD. Neuraxial anesthesia (NA) is the preferred anesthetic for CD because it has a better safety profile, avoids airway management, decreases blood loss, improves postoperative analgesia, and decreases neonatal drug exposure compared with general anesthesia.

NA allows the patient and partner to experience the delivery, enhancing parent-baby bonding, but has many well-described risks, including hypotension leading to nausea, shivering, post-dural puncture headache, nerve injury, and failure to achieve satisfactory anesthesia. If a CD is needed in a parturient with an existing labour epidural analgesia, it is common practice to convert or 'top-up' the epidural catheter, with the aim of initiating surgical anesthesia by injecting more concentrated local anesthetic (LA) solution, normally combined with a lipid-soluble opioid.

Patients' greatest concern during and after CD is pain. Childbirth is a profound experience with 1/3 of patients experiencing a highly stressful and potentially traumatic childbirth. A birthing parent's experience during a planned CD versus an unexpected CD (uCD) can play a role in the development of post-traumatic stress disorder (PTSD). Childbirth-related PTSD is estimated to affect 5-6% of all postpartum women. With CD representing 1/3 of all North American deliveries annually, uCDs will contribute to an increased risk of PTSD and post-partum depression (PPD) symptoms. Given the suffering associated with PPD and that women experiencing PPD incur greater health care costs, understanding the association between CD and associated traumatic birth experiences may help guide interventions to address both the psychosocial impact on families and the economic impacts on health care.

The concept of "patients as educators" is new to the practice of anesthesia and aims to embrace the patient perspective to guide quality improvement initiatives. This study will explore patients' perception of their experience with uCD under neuraxial anesthesia (uCD-NA) and aim to provide insight into patients' feelings, concerns and expectations after an unscheduled experience for childbirth. By adding the providers' perspective on the topic of childbirth via uCD-NA, the investigators will be able to explore differences and similarities in opinions, thoughts, feelings and concerns as well as wishes for their care between patients and their providers. Thus, the study will also aim to explore the perspective of anesthesiologists, anesthesia assistants/respiratory therapists, obstetricians and registered nurses.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* English language proficiency (as interviews will be performed in English)
* ASA Physical Classification Score 2-5 +/- E
* Emergency or Urgent CD that can be done with the existing or newly applied neuraxial anesthesia (specifically, without the need for general anesthesia) due to fetal or maternal emergencies (e.g., fetal bradycardia, pre-eclampsia, chorioamnionitis, etc.)
* uCD is defined as Level 1 (Emergency - Immediate threat to life of woman or fetus) and Level 2 (Urgent - Maternal or fetal compromise which is not immediately life-threatening) CD 16
* Patients will be included if they undergo preterm delivery (under 37 weeks of gestation, or are having a multiple gestation pregnancy, also, if there is a significant fetal anomaly present

Exclusion criteria:

* Under 18 years of age
* Unable to answer questions due to a language barrier or because of their mental or physical state (e.g., intubated patients)
* BMI at the time of delivery that falls in the super-morbidly obese category (BMI > 55 kg/m2)
* Patients who underwent preterm delivery (under 32 weeks gestation)
* Patients will be excluded if neonatal death has occurred.
* Patients who were scheduled for an elective CD will be excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who deliver by unexpected cesarean section with neuraxial anesthesia at Mount Sinai Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Patient questionnaire | Following cesarean delivery, and prior to hospital discharge (at approximately 48 hours postpartum).
  Patients will be asked to rate their experience of having a cesarean delivery with neuraxial anesthesia, in terms of satisfaction and their experience with any discomfort. Some questions are yes/no, some are on a scale from 1-10, where 1 = not at all and 10 = totally agree, and some are open-ended. The questionnaire will take approximately 10 minutes to complete.
Patient interview | Following cesarean delivery, and prior to hospital discharge (at approximately 48 hours postpartum).
  Patients will be interviewed in person by a member of the research team and asked open ended questions. Interviews will be recorded, transcribed and coded for themes. Responses are not reported on any scale. The interview will take approximately 30 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Nabecker, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No